CLINICAL TRIAL: NCT04647448
Title: Multisensor Array for the Localisation of Coronary Artery Stenosis
Brief Title: Multisensor Array for the Localisation of Coronary Artery Stenosis (MALCAS)
Acronym: MALCAS
Status: Withdrawn | Type: Observational
Why Stopped: Abandoned
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: Imperial College London (Other); Brunel University (Other)
Responsible Party: Sponsor
Other Study IDs: 274197
Record Dates: First submitted 2020-07-27; First posted 2020-12-01 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: CORONARY ARTERY DISEASE
Keywords: Phono-cardiography
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy volunteers: Participants with no known cardiovascular disease
  Interventions: Diagnostic Test: Application of sensor patch
- Chest pain: Patients with symptoms of chest pain, undergoing elective coronary artery CT
  Interventions: Diagnostic Test: Application of sensor patch

INTERVENTIONS:
Diagnostic Test: Application of sensor patch — Application of sensor patch to chest to record acoustic signals due to disturbed blood flow.

SUMMARY:
This is a proof of concept study involving a novel medical device, developed to investigate the potential for detecting and localising coronary artery stenosis. A prototype device will be used in the proposed clinical investigation. It is a stick-on patch containing sensors which measure the sound produced at and the movement of, the chest surface by flowing blood as it accelerates through the stenosis and becomes disturbed as it emerges downstream, allowing the blockage to be detected and localised non-invasively.

The proposed clinical investigation will involve a small number of patients and healthy volunteers. The patients will be drawn from those attending The BartsHeart Centre for suspected or diagnosed coronary artery disease and all clinical measurements will take place at Barts Health Trust. The patch to be used in the proposed clinical investigation incorporates commercially available sensors and will be tested by recording acoustic signatures in healthy volunteers, then in patients undergoing coronary CT angiography at Barts. Signals will be analysed initially by measuring their acoustic energy at various frequencies and in later iterations, by a machine-learning algorithm. Results will be validated against the CT angiography gold standard.

DETAILED DESCRIPTION:
This project is a trial of a novel device, in the form of a stick-on patch containing miniature accelerometers and microphones, designed to detect sounds produced by disturbed blood flow in stenosed coronary arteries. Initially, acoustic data will be collected from a small group of healthy volunteers to confirm proof of concept. Recordings from the patch will then be made on up to 100 patients who, having presented with chest pain to the Barts Heart Clinic, are undergoing simultaneous CTa investigations to determine the presence or absence of occlusive CAD.

The purpose of the study is to determine if the nature of the signals recorded by the patch makes it possible to distinguish those patients who have identifiable CAD, as detected by CTa (the reference method) from those in whom no occlusive lesions can be seen in the CTa images. The measurements on patients will be preceded by a trial on 20 healthy volunteers to establish base line readings and to ensure the reliability of the patch and the associated data acquisition system, in the field.

Coronary artery disease (CAD) is the leading cause of death worldwide. In Europe alone in 2014 the resulting cost of health care, and lost production was around €100 billion per year. Existing diagnostic methods apart from ECG require skilled operators and expensive equipment.

Recent advances in cCTA make it possible to detect and localise occlusive lesions with high accuracy and precision, whilst minimising the use of contrast media, albeit at the cost of some exposure to ionising radiation. Of equal or greater concern is the fact that approximately 2/3 of symptomatic patients are found, on investigation, to be occlusion-free, representing a great waste of resources and thus a loss of productivity for the healthcare system and the patients themselves, to say nothing of their distress on facing a false positive diagnosis and the risks associated with contrast injection and exposure to unnecessary ionising radiation.

The non-invasive system proposed here would be applied to symptomatic patients with stable chest pain attending a cardiac outpatient clinic with the intention of screening out the 2/3 mentioned above, resulting in large cost and time savings.

More generally, prevention of CAD, facilitated by routine screening in a primary care setting would also have the potential to relieve the economy of a major burden. Thus, there is scope for enormous life and cost saving in the early-days detection and mitigation of CHD. Apart from the immediate cost savings the longer term benefits include, for example, more appropriate allocation of imaging infrastructure, streamlining of patients in intermediate risk categories who require a more refined risk stratification; a novel technology with potential application to other near surface sites (e.g. carotid stenosis) and with potential development for deep sites (e.g. femoral stenosis); a sensing device suited to the localisation software being developed by co-workers arising from our previous EPSRC funding. There is also the potential for a 'take home' diagnostic kit which can collect and report data via domestic WiFi.

Current assessment of patients with symptoms of CAD who are referred to cardiac clinics is in most cases recommendation for a non-invasive imaging test, followed, if positive, by invasive coronary angiography. In 2010-2012 at Barts Health only 25% of coronary CT angiography scans were followed by invasive confirmation of advanced disease or treatment with either coronary angioplasty or bypass graft surgery. This was observed in a population of patients "appropriately referred" to testing, according to current NICE clinical guideline 95.

This percentage is in keeping with a large US multicentre registry where around 65% of the patients were found to be free of occlusive vascular disease following angiographic investigation. This study also showed that, although some demographic and clinical characteristics could be useful in determining the likelihood of obstructive coronary artery disease, the incremental value of non-invasive tests (resting ECG, echocardiography, imaging stress tests and coronary CT angiography) was limited. The implications are two-fold: whilst clinical assessment alone is insufficient to diagnose or exclude the presence of disease, imaging tests have an exceedingly low diagnostic yield. It was estimated that the volume of unnecessary non-invasive tests performed in the US in the decade between 2000 and 2010 cost the US economy more than $500m.

Despite impressive technological advances in medical imaging equipment introduced over the last years, translating into better accuracy and precision, we are witnessing a paradoxical increase in the number of imaging tests performed per year, which also includes multiple testing in the same patient .

Given the financial pressure on the healthcare system, large numbers of unnecessary imaging tests are unsustainable, as are the productivity losses related to hospital visits, the risks of false positive findings, and unnecessary referrals to invasive procedures which expose patients to the risk of complications (e.g. bleeding, contrast induced nephropathy, stroke, repeat radiation exposure).

The investigators propose a non-invasive system to pre-screen symptomatic patients attending a cardiac outpatients' clinic. This approach is aimed at supporting a more appropriate use of imaging resources, refining the identification of patients requiring an imaging test and/or an invasive procedure, reducing the number of unnecessary imaging tests and angiographic investigations, resulting in large cost and time savings.

ELIGIBILITY:
Inclusion Criteria (healthy volunteers):

* Healthy
* Not pregnant

Inclusion Criteria (patients):

* Presenting with chest pain with possibility of coronary artery disease
* No infectious disease or neoplasia

Exclusion Criteria (healthy volunteers):

* Considered by the study clinician to be unsuitable to participate
* Considered by the clinical research team to be incapable of providing written informed consent for any reason.

Exclusion Criteria (patients):

* Considered by the clinical research team to be incapable of providing written informed consent for any reason.
* Considered by their healthcare professional to be unsuitable to participate
* Participation in another ongoing drug or medical device study
* Participation in a drug study within the 3 months prior to the date of potential enrolment into this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male and female, minimum age 18 years. Healthy volunteers selected by advertisement Patients selected from those attending Barts Heart Centre for elective coronary CT angiography.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy | Through study completion, 1 year
  Diagnostic accuracy of the device (stick-on patch) for indicating the presence or absence of one or more coronary arterial stenoses as indicated by the reference method (CT angiography results)

SECONDARY OUTCOMES:
Stenosis severity | Through study completion, 1 year
  Comparison of the magnitude of the disturbed flow to the severity of the stenosis as measured from the CTa images.
Number of stenoses | Through study completion, 1 year
  To determine agreement between the number of stenoses detected by the reference method and the number suggested by the signal characteristics of the test device
Stenosis position | Through study completion, 1 year
  To assess the degree of agreement between the position of each stenosis as determined by the reference method and the position suggested by the signal characteristics of the test device

IPD SHARING:
Plan to Share IPD: No
IPD to be shared with named collaborators for further analysis.

REFERENCES:
- [Background] Andrus BW, Welch HG. Medicare services provided by cardiologists in the United States: 1999-2008. Circ Cardiovasc Qual Outcomes. 2012 Jan;5(1):31-6. doi: 10.1161/CIRCOUTCOMES.111.961813. Epub 2012 Jan 10. PMID 22235064
- [Background] Ladapo JA, Blecker S, Douglas PS. Physician decision making and trends in the use of cardiac stress testing in the United States: an analysis of repeated cross-sectional data. Ann Intern Med. 2014 Oct 7;161(7):482-90. doi: 10.7326/M14-0296. PMID 25285541
- [Background] Nichols M, Townsend N, Scarborough P, Rayner M. Cardiovascular disease in Europe 2014: epidemiological update. Eur Heart J. 2014 Nov 7;35(42):2950-9. doi: 10.1093/eurheartj/ehu299. Epub 2014 Aug 19. PMID 25139896
- [Background] Patel MR, Peterson ED, Dai D, Brennan JM, Redberg RF, Anderson HV, Brindis RG, Douglas PS. Low diagnostic yield of elective coronary angiography. N Engl J Med. 2010 Mar 11;362(10):886-95. doi: 10.1056/NEJMoa0907272. PMID 20220183
- [Background] Villadsen PR, Petersen SE, Dey D, Zou L, Patel S, Naderi H, Gruszczynska K, Baron J, Davies LC, Wragg A, Botker HE, Pugliese F. Coronary atherosclerotic plaque burden and composition by CT angiography in Caucasian and South Asian patients with stable chest pain. Eur Heart J Cardiovasc Imaging. 2017 May 1;18(5):556-567. doi: 10.1093/ehjci/jew085. PMID 27225816